CLINICAL TRIAL: NCT05242393
Title: The Role of Circadian Factors in Regulation of Neuroplasticity in Ischemic Stroke (Observational)
Status: Recruiting | Type: Observational
Sponsor: Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health (Other)
Responsible Party: Principal Investigator, Lyudmila Korostovtseva, Senior Researcher, Department for Hypertension, Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health
Other Study IDs: 21-75-1017-2 (observational)
Record Dates: First submitted 2022-01-26; First posted 2022-02-16 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Stroke, Ischemic; Sleep Disorder
Keywords: neuroplasticity; cognitive dysfunction; disability; circadian rhythm; functional deficit; stroke outcome; sleep-disordered breathing; heart rate variability
MeSH Terms: conditions — Ischemic Stroke; Sleep Wake Disorders; Cognitive Dysfunction; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — whole blood, serum, saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Retrospective cohort: Patients with acute ischemic stroke admitted to the Stroke Unit of one participating center in 2018-2022. The data collected within clinical routine will be analyzed including stroke characteristics at baseline and at discharge (10-14 days after admission), neuroimaging data, sleep characteristics (routine polygraphy study), heart rate variability, routine blood tests.
  Interventions: Other: No intervention is planned
- Prospective cohort: Approximately 200-250 patients with acute ischemic stroke admitted to the Stroke Unit of one participating center in 2022-2024 will undergo the assessment of medical records, stroke characteristics, the assessment of sleep characteristics and blood sampling for the evaluation of genetic biomarkers of circadian rhythms at baseline (within 2-3 days of admission) and at 10-14 days (at discharge).
  Interventions: Other: No intervention is planned

INTERVENTIONS:
Other: No intervention is planned — No intervention is planned

SUMMARY:
The study is aimed at the investigation of the association of biomarkers of circadian rhythms with sleep characteristics and stroke outcome in acute stroke patients. It is designed as an observational cohort study with the retrospective and prospective longitudinal arms.

DETAILED DESCRIPTION:
In the retrospective arm of the study, the routinely collected data of patients admitted to the stroke unit with acute ischemic stroke (from 2018 till 2022) will be evaluated. In the prospective longitudinal arm, about 200-250 patients admitted to the Stroke Unit of one participating center will undergo examination including the assessment of medical records, stroke characteristics, sleep characteristics and blood sampling for the evaluation of genetic biomarkers of circadian rhythms within the first 2-3 days after admission.The assessment of stroke severity and functional deficit will be repeated at 10-14 days after stroke.

The following associations will be assessed:

* the association of genetic biomarkers of circadian rhythms with stroke outcome (the difference in neurological and functional deficit from admission to 14th day after stroke), with stroke characteristics (stroke subtype and neuroimaging stroke parameters) and with sleep characteristics.
* the association of sleep characteristics with stroke outcome (the difference in neurological and functional deficit from admission to 14th day after stroke) and with stroke characteristics (stroke subtype and neuroimaging stroke parameters).

ELIGIBILITY:
Inclusion Criteria:

* acute (symptom onset to admission <1 days) ischemic stroke
* ischemic stroke affecting the branches of anterior cerebral artery, middle cerebral artery and posterior cerebral artery
* age 18-80 years
* moderate or severe stroke (National Institutes of Health Stroke Scale, NIHSS>=5)
* intravascular stroke treatment with thrombolysis or thrombectomy leading to satisfactory reperfusion (if applicable)
* informed consent

Exclusion Criteria:

* secondary parenchymal hemorrhage (>hemorrhage index -2)
* clinically unstable or life-threatening conditions
* known progressive neurological diseases
* known psychiatric diseases
* concomitant benzodiazepine medication
* drug or alcohol abuse
* pregnancy
* disability to participate in the study
* congestive heart failure with reduced ejection fraction (<=45%) or New York Heart Association (NYHA) classification III-IV functional class

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the patients with confirmed acute ischemic stroke admitted to the Stroke Unit
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the value of National Institutes of Health Stroke Scale from baseline to 14th day after inclusion | From baseline to 14th day after treatment initiation
  National Institutes of Health Stroke Scale (NIHSS) is a tool used to objectively quantify the impairment caused by a stroke, 0-42 scores, higher scores characterize worse impairment
Stroke-related disability assessed by the change in modified Rankin scale from baseline to 14th day after treatment initiation | From baseline to 14th day after treatment initiation
  values of modified Rankin scale (scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke, from 0 (no symptoms) to 6 (dead) points)
Stroke-related disability assessed by the change in Rivermead Mobility Index from baseline to 14th day after treatment initiation | From baseline to 14th day after treatment initiation
  a standardized scale used to assess mobility in patients with neurological deficits, a maximum of 15 points is possible; higher scores indicate better mobility performance
Stroke-related disability assessed by the change in Barthel Index from baseline to 14th day after treatment initiation | From baseline to 14th day after treatment initiation
  a common scale used to measure performance in activities of daily living, 0-100 scores, higher scores define better performance

SECONDARY OUTCOMES:
Sleep quality assessed by Pittsburgh Sleep Quality Index | Baseline
  Pittsburgh Sleep Quality Index is a self-rated questionnaire which assesses sleep quality and disturbances over the last (previous) 1-month (a retrospective assessment) time interval, Each of the sleep components yields a score ranging from 0 to 3, with 3 indicating the greatest dysfunction. The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score indicating worse sleep quality
Sleepiness assessed by Epworth Sleepiness Scale | Baseline
  a common tool to assess sleepiness; 0-24 points, higher score indicate greater sleepiness
Fatigue assessed by Fatigue severity Scale | Baseline
  a common 9-item tool used to determine and quantify fatigue as subjective feeling of exhaustion, persisting lack of energy and rapid inanition, 9-63 points, higher score indicates more severe fatigue
Insomnia assessed by Insomnia severity index | Baseline
  a 7-item tool to assess the severity of insomnia, 0-5 points per each item, higher score indicates more severe insomnia
Chronotype assessed by Morningness-Eveningness Questionnaire | Baseline
  a common 19-item tool to estimate individual chronotype, a score ranging from 16 to 86; scores of 41 and below indicate "evening types", scores of 59 and above indicate "morning types", scores between 42-58 indicate "intermediate types"

OTHER OUTCOMES:
sleep-related respiratory characteristics: apnea-hypopnea index | Baseline
  assessed by routine polygraphy: apnea-hypopnea index (higher values indicate greater severity; <5 episodes/h - normal, >=5 episodes/h - pathological)
sleep-related respiratory characteristics: oxygen desaturation index | Baseline
  assessed by routine polygraphy: oxygen desaturation index (higher values indicate greater severity; <5 episodes/h - normal, >=5 episodes/h - pathological)
sleep-related respiratory characteristics: time under oxygen saturation <90% | Baseline
  assessed by routine polygraphy: time under oxygen saturation <90% (higher values indicate greater severity), in minutes
sleep-related respiratory characteristics: average oxygen saturation | Baseline
  assessed by routine polygraphy: average oxygen saturation (lower values indicate greater severity), in %
sleep-related respiratory characteristics: lowest oxygen saturation | Baseline
  assessed by routine polygraphy: lowes oxygen saturation (lower values indicate greater severity), in %
Nocturnal heart rate variability characteristics derived from nocturnal pulseoximeter data: standard deviation of normal-to-normal intervals | Baseline
  standard deviation of normal-to-normal intervals (msec)
Nocturnal heart rate variability characteristics derived from nocturnal pulseoximeter data: number of interval differences of successive heart beats greater than 50 ms | Baseline
  number of interval differences of successive heart beats greater than 50 ms
Nocturnal heart rate variability characteristics derived from nocturnal pulseoximeter data: spectral power in high-frequency power bands | Baseline
  spectral power in high-frequency power bands (Hz)
Nocturnal heart rate variability characteristics derived from nocturnal pulseoximeter data: spectral power in low-frequency power bands | Baseline
  spectral power in low-frequency power bands (Hz)
Sleep duration assessed by polysomnography | Baseline
  Sleep duration (minutes)
Sleep efficiency assessed by polysomnography | Baseline
  sleep efficiency (%)
Sleep latency assessed by polysomnography | Baseline
  sleep latency (minutes)
Sleep S1 stage duration assessed by polysomnography | Baseline
  S1 sleep stage percentage of total sleep time (%)
Sleep S2 stage duration assessed by polysomnography | Baseline
  S2 sleep stage percentage of total sleep time (%)
Sleep S3 stage duration assessed by polysomnography | Baseline
  S3 sleep stage percentage of total sleep time (%)
Rapid eye movement (REM) stage duration assessed by polysomnography | Baseline
  Rapid eye movement (REM) sleep stage percentage of total sleep time (%)
Wake after sleep onset time assessed by polysomnography | Baseline
  wake after sleep onset time (minutes), higher values indicate worse disturbance
Arousal index assessed by polysomnography | Baseline
  Arousal index (episodes/hour of sleep), higher values indicate worse disturbance
periodic limb movement index assessed by polysomnography | Baseline
  periodic limb movement index (episodes/hour of sleep), higher values indicate worse disturbance
Stroke lesion volume | Baseline
  Stroke lesion volume assessed by neuroimaging (computer tomography scan or magnetic resonance imaging) (ml or mm3)

CONTACTS AND LOCATIONS:
Overall Officials: Lyudmila Korostovtseva, MD, PhD, Principal Investigator — Almazov National Medical Research Centre
Locations (1):
- Almazov National Medical Research Centre, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Korostovtseva L. Ischemic Stroke and Sleep: The Linking Genetic Factors. Cardiol Ther. 2021 Dec;10(2):349-375. doi: 10.1007/s40119-021-00231-9. Epub 2021 Jun 30. PMID 34191267
- [Background] Bochkarev MV, Korostovtseva LS, Medvedeva EA, Rotar OP, Sviryaev YV, Zhernakova YV, Shalnova SA, Konradi AO, Chazova IE, Boitsov SA, Shlyakhto EV. [Sleep disorders and stroke: data of the esse-rf study]. Zh Nevrol Psikhiatr Im S S Korsakova. 2019;119(4. Vyp. 2):73-80. doi: 10.17116/jnevro201911904273. Russian. PMID 31317919
- [Background] Seiler A, Camilo M, Korostovtseva L, Haynes AG, Brill AK, Horvath T, Egger M, Bassetti CL. Prevalence of sleep-disordered breathing after stroke and TIA: A meta-analysis. Neurology. 2019 Feb 12;92(7):e648-e654. doi: 10.1212/WNL.0000000000006904. Epub 2019 Jan 11. PMID 30635478